CLINICAL TRIAL: NCT03256175
Title: The Effects Of Peri-Percutaneous Coronary Intervention Oxygenation On Myocardial Protection And Cardiovascular Function: A Pilot Study
Brief Title: The Effect of Peri-percutaneous Coronary Intervention Oxygenation on Myocardial Protection & Cardiovascular Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1198.49
Record Dates: First submitted 2017-07-31; First posted 2017-08-21 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Ischemia; Cardiovascular Morbidity
Keywords: Myocardial Protection; Oxygen; Exercise Test
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both medical air and oxygen were supplied in compressed liquid form and available throughout the hospital. During the study, the medical gas cylinders shielded using an opaque temporary cover. Similarly the oxygen saturation was not displayed, but instead monitored by an independent third party.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen (Experimental): Patient was give 15L/min of Oxygen via HFM 30 mins before and continue through out the procedure. 6 weeks post procedure, EST was arranged
  Interventions: Procedure: Percutaneous Coronary Intervention
- Air (Placebo Comparator): Patient was given Facemask without oxygen through out the procedure. 6 weeks post procedure, EST was arranged
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — PCI technique (e.g. pre-dilatation vs. direct stenting and stent choice) was left to operator discretion. Stent post dilatation was permitted as per individual operator practice

SUMMARY:
Elective percutaneous coronary intervention (PCI) is often associated with myocardial necrosis evidenced by peri-procedural troponin release. This is a surrogate for subsequent cardiovascular events. There is no study on the effect of peri-PCI oxygenation in in myocardial protection and cardiopulmonary fitness outcome. Patients with higher baseline cardiopulmonary fitness will have lower mortality.

This study is to assess the utility of oxygen to reduce ischaemia in patients with significant stable coronary artery disease scheduled for elective PCI. The secondary objective is to evaluate further effect of peri- PCI oxygenation on cardiovascular fitness and autonomic response.

DETAILED DESCRIPTION:
OBJECTIVE: This study is to assess the utility of oxygen to reduce ischaemia in patients with significant stable coronary artery disease scheduled for elective PCI. The secondary objective is to evaluate further effect of peri- PCI oxygenation on cardiovascular fitness and autonomic response.

STUDY DESIGN: Randomized double blinded prospective pilot study SAMPLE SIZE: 30 patients scheduled for elective for PCI randomized to 2 groups, oxygen group ( 15L/min) and air group METHOD: Patient whom fulfil inclusion criteria were recruited and randomized to 2 groups via computer allocation system. The assigned inhaled gas will be delivered via high-flow mask at 15L/min for a minimum of 30 minutes immediately prior to and continued throughout the PCI procedure. Patients were blinded throughout the procedure but the practising cardiologist and staff nurses were not blinded. Routine care continued post PCI. Blood sampling for Troponin I was taken at 6 hours and 24 hours following stent implantation. Patients were discharged one day after the procedure as per current routine practice.

Patients were given routine follow up with the cardiac rehabilitation clinic in 4 weeks time post discharge. EST was arranged 6 weeks post procedure PRIMARY OUTCOME MEASURE: Troponin I at 6 and 24 hours SECONDARY OUTCOME MEASURE: METs, Heart Rate Recovery, Chronotropic Index

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Haemodynamically important coronary artery disease (>70% luminal stenosis angiographically in ≥1 major epicardial coronary artery

Exclusion Criteria:

* Significant chronic airways disease with type-2 respiratory failure precluding safe use of oxygen
* Coronary stenoses where evidence of plaque instability is evident e.g. rest pain, visual evidence of thrombus, elevation of Troponin T at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess the myocardial protection | 6 hours and 24 hours after the procedure
  this is done by comparing changes Troponin I at 6 (baseline) to 24 hours between both study arms.

SECONDARY OUTCOMES:
To assess the utility of peri-PCI oxygenation to improve cardiovascular fitness | 6 weeks post procedure
  assessed by Functional capacity in METs-Maximum METs achieved
To assess the utility of peri-PCI oxygenation to improve autonomic response | 6 weeks post procedure
  assessed by Heart Rate Recovery
To assess the utility of peri-PCI oxygenation to improve autonomic response | 6 weeks post procedure
  assessed by Chronotropic Index

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Chan, MBBS, Principal Investigator — schin1022@yahoo.com; Anwar Suhami, MBBS, Study Chair — anwar@ummc.edu.my

IPD SHARING:
Plan to Share IPD: Undecided